CLINICAL TRIAL: NCT00189501
Title: A Multi-Center, Observational Registry of Subjects With Secondary Hyperparathyroidism (HPT) and Chronic Kidney Disease (CKD)
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Other Study IDs: 20040159
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Nephrology
Keywords: Chronic Kidney Disease, CKD,; Secondary Hyperparathyroidism, HPT
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary | interventions — Cinacalcet

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Sensipar®

SUMMARY:
Objectives include description of current practices; assessment over time of K/DOQI goals, clinical outcomes, health resource utilization(HRU) and patient reported outcomes (PRO) and the impact of Sensipar® on these parameters

ELIGIBILITY:
Inclusion Criteria:

* 3 month history of Stage 4 or Stage 5 CKD
* A PTH value within 3 months of enrollment
* If relevant, completion of Sensipar® study prior to enrolling in Registry Exclusion Criteria:
* Females who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com